CLINICAL TRIAL: NCT02640859
Title: Investigation of Metabolic Risk in Korean Adults
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-Biobank
Record Dates: First submitted 2015-12-19; First posted 2015-12-29 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — For measuring biomarkers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal cohort: Normal cohort for biobank

SUMMARY:
A cohort study with Korean adults to investigate biomarkers in prediction of cardiometabolic and other diseases

DETAILED DESCRIPTION:
This is a prospective cohort study with Korean adults to investigate biomarkers in prediction of cardiometabolic and other diseases

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without chronic diseases
* Diabetic patients who are well controlled with oral antidiabetic agents
* Hypertensive patients who are well controlled with oral antihypertensive agents
* Dyslipidemic patients who are well controlled with oral lipid-lowering agents

Exclusion Criteria:

* Malignancy
* Chronic wasting disease
* Long-term steroid use

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Korean Adults
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiovascular disease | 5 years

SECONDARY OUTCOMES:
Incidence of diabetes mellitus | 5 years
Incidence of fatty liver | 5 years
Incidence of metabolic syndrome | 5 years
Incidence of osteoporosis | 5 years
Incidence of sarcopenia | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, PhD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No